CLINICAL TRIAL: NCT03918499
Title: A Phase 1b/2 Trial of the IRX-2 Regimen and Pembrolizumab in Patients With Advanced Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: IRX-2, Cyclophosphamide, and Pembrolizumab in Treating Participants With Recurrent or Metastatic Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18069; NCI-2018-01885 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18069 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2018-09-10; First posted 2019-04-17 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Recurrent Gastric Adenocarcinoma; Recurrent Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Cyclophosphamide; IRX 2; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, cyclophosphamide, and IRX-2) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1. Participants also receive cyclophosphamide IV on day 1 and IRX-2 SC for 10 days starting on day 4 during cycles 1, 5, 9, 13, 17, 21, 25, 29, and 33. Treatment repeats every 3 weeks for up to 35 cycles in the absence of disease or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Cytokine-based Biologic Agent IRX-2; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Cytokine-based Biologic Agent IRX-2 — Given SC
  Other Names: IRX-2
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase Ib/II trial studies the side effects of IRX-2, cyclophosphamide, and pembrolizumab work in treating participants with gastric or gastroesophageal junction cancer that has come back or that has spread to other places in the body. Interleukins, such as those found in IRX-2, are proteins made by white blood cells and other cells in the body and may help regulate immune response. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving RX-2, cyclophosphamide, and pembrolizumab may work better in treating participants with gastric or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of combination IRX-2 regimen and pembrolizumab.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate of IRX-2 regimen combined with pembrolizumab using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune modified RECIST criteria.

II. To evaluate initial median progression-free and overall survival in these patients treated with combination IRX-2 regimen and pembrolizumab.

EXPLORATORY OBJECTIVES:

I. To evaluate the circulating T cell profiles in patients before and after therapy with combination IRX-2 regimen and pembrolizumab.

II. To evaluate the baseline and post-treatment tumor tissue immune gene expression profiling using the Nanostring platform.

III. To explore identification of tumor tissue neoantigens through a multiplex proteomic assay (MHC-PepSeq) paired with tumor genomic and transcriptomic sequencing.

IV. To explore putative biomarkers (including circulating tumor deoxyribonucleic acid [DNA] and immune cell profiles) in peripheral blood to generate hypotheses for response to treatment with combination IRX-2 regimen and pembrolizumab.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Participants also receive cyclophosphamide IV on day 1 and IRX-2 subcutaneously (SC) for 10 days starting on day 4 during cycles 1, 5, 9, 13, 17, 21, 25, 29, and 33. Treatment repeats every 3 weeks for up to 35 cycles in the absence of disease or unacceptable toxicity.

After completion of study treatment, participants are followed up for 30 days and then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed recurrent or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma progressed or intolerant to >= 2 lines of systemic therapy.
* Patients must have recurrent or metastatic gastric/GEJ adenocarcinoma that are not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
* Willing and able to give informed consent and adhere to protocol therapy; written informed consent and any locally required authorization must be obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
* No prior exposure to PD-1/PD-L 1 inhibitor therapy.
* Patients are deemed eligible for pembrolizumab therapy with tumors demonstrating PD-L1 expression by the Combined Positive Score (CPS) being >= 1 as per the Food and Drug Administration (FDA)-approved Dako PD-L1 immunohistochemistry (IHC) 22C3 PharmDx assay.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* Body weight must be > 30 Kg.
* Hemoglobin > 8 g/dL.
* Absolute neutrophil count (ANC) > 1,200 x 10^9/mL.
* Platelet count > 75 x 10^9/mL.
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) OR direct bilirubin =< ULN if total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/serum glutamate-pyruvate transaminase [SGPT]) =< 5 x ULN.
* Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.5 x the ULN.
* Serum creatinine =< 1.5 x ULN OR measured creatinine clearance (CL) > 40 mL/min or calculated creatinine clearance CL > 40 mL/min by the Cockcroft-Gault formula or by 24- hour urine collection for determination of creatinine clearance.
* Palliative radiation therapy is allowed to non-target lesions at the discretion of the treating physician.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) or evaluable disease as outlined in Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Life expectancy of greater than 3 months in the opinion of the treating physician.
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Prior exposure to the IRX-2 regimen and/or PD-1/PD-L1 inhibitors are excluded.
* Radiation therapy with a curable intent within 30 days of first dose of study treatment is excluded. However, radiation therapy with a palliative intent is allowed as long as treatment with study medication occurs >= 14 days after the last dose of radiation.
* Any medical contraindications or previous therapy that would preclude treatment with the IRX-2 regimen or pembrolizumab.
* Known allergies to ciprofloxacin or phytohemagglutin given trace amount of these agents are contained in IRX-2.
* Patients with ongoing chronic myelosuppression, myelodysplasia, or hemorrhagic cystitis which would contraindicate receipt of cyclophosphamide.
* Any unresolved toxicity National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with IRX-2, pembrolizumab may be included only after consultation with the study physician.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia.
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients without active disease in the last 2 years may be included but only after consultation with the study physician.
  * Patients with celiac disease controlled by diet alone.
* Current or prior use of immunosuppressive medication within 14 days prior to cycle 1, day 1. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroid or local steroid injections (e.g., intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
* Major surgical procedure (as defined by the Investigator) within 28 days prior to cycle 1, day 1. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogeneic organ transplantation.
* Symptomatic cardiopulmonary disease (including congestive heart failure and hypertension), coronary artery disease, serious arrhythmia or chronic lung disease. Patients with these conditions who are stable with relatively minor symptoms and who are appropriate candidates for systemic treatments need not be excluded.
* Myocardial infarction within the last 3 months.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has a history of active hepatitis B requiring ongoing antiviral therapy or a history of untreated hepatitis C.
* Has received a live vaccine within 4 months of planned start of study therapy (cycle 1, day 1).

  * Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed provided not within 4 weeks of planned start of study therapy (cycle 1, day 1); however intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed.
* Signs or symptoms of systemic infection (use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection).
* Stroke or other symptoms of cerebral vascular insufficiency within the last 3 months.
* Previous diagnosis of invasive cancer from which the individual is not disease-free AND that has required treatment within the past 3 years, except for superficial skin, cervical cancer in-situ, or early stage prostate or bladder cancer (i.e. treatment with curative intent and long term disease-free expectations).
* History of leptomeningeal carcinomatosis.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to one year after last dose of cyclophosphamide or 180 days after the last dose of pembrolizumab therapy, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chao, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2): Participants receive 200 mg of pembrolizumab IV over 30 minutes on day 1. Participants also receive 300 mg/m2 of cyclophosphamide IV on day 1 and 230 or 460 units of IRX-2 SC for 10 days starting on day 4 during cycles 1, 5, 9, 13, 17, 21, 25, 29, and 33. Treatment repeats every 3 weeks for up to 35 cycles in the absence of disease or unacceptable toxicity.
  IRX-2 is supplied as a pale yellow, sterile liquid for subcutaneous injection in a 2.0 ml single dose vial.
  Cyclophosphamide: Given IV
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Hispanic | 2
  Non-Hispanic White | 4
Region of Enrollment [Number; unit: participants]
  United States | 9
Tumor Stage @ Diagnosis [Count of Participants; unit: Participants] — Stage I-III: Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV: The cancer has spread to distant parts of the body.
  Participants
    II | 2
    IV | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From initial treatment until progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first day of study drug administration to disease progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
Number analyzed (Participants) | 9
Months | 1.1 [0.4 to 2.0]

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From the time of initial treatment until death from any cause.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
Number analyzed (Participants) | 9
Months | 2.9 [0.4 to 8.7]

3. Secondary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years and 6 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2)
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2) (N=9)
Pericardial effusion (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Cyclophosphamide, and IRX-2) (N=9)
Anemia (Blood and lymphatic system disorders) | 9 (24)
Atrial fibrillation (Cardiac disorders) | 1 (4)
Palpitations (Cardiac disorders) | 1 (4)
Pericardial effusion (Cardiac disorders) | 1 (4)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Tricuspid valve disease (Cardiac disorders) | 1 (4)
Mitral valve disease (Cardiac disorders) | 1 (4)
Pulmonary valve disease (Cardiac disorders) | 1 (4)
Aortic valve disease (Cardiac disorders) | 1 (4)
Abnormal QRS-T angle, consider primary T (Cardiac disorders) | 1 (2)
Non-specific T Wave Abnormality (Cardiac disorders) | 1 (1)
ST and T Wave Abnormality (Cardiac disorders) | 1 (3)
Sinus Bradycardia (Cardiac disorders) | 1 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
T Wave Abnormality (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
10005886-Blurred vision (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (3)
Double Vision (Eye disorders) | 1 (4)
Double vision (Eye disorders) | 1 (1)
Retinal Hemorrhage (Eye disorders) | 1 (5)
Swelling around the eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (13)
Ascites (Gastrointestinal disorders) | 2 (4)
Bloating (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 5 (15)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 5 (13)
Nausea (Gastrointestinal disorders) | 7 (12)
Vomiting (Gastrointestinal disorders) | 4 (12)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4)
Acid Reflux (Gastrointestinal disorders) | 1 (3)
Early Satiety (Gastrointestinal disorders) | 1 (3)
Teeth Sensitivity (Gastrointestinal disorders) | 1 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (26)
Fever (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 1 (2)
Pain (General disorders) | 3 (12)
Edema limbs (General disorders) | 3 (9)
Non-cardiac chest pain (General disorders) | 1 (2)
Left Lower Extremity Edema (General disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (3)
Activated partial thromboplasti (Investigations) | 1 (4)
Alanine aminotransferase increa (Investigations) | 2 (6)
Alkaline phosphatase increased (Investigations) | 7 (23)
Aspartate aminotransferase incr (Investigations) | 2 (8)
Blood bilirubin increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (7)
Thyroid stimulating hormone inc (Investigations) | 3 (10)
White blood cell decreased (Investigations) | 1 (1)
Hyperchloremia (Investigations) | 2 (3)
Hypochloremia (Investigations) | 1 (1)
Hypochlorinemia (Investigations) | 2 (4)
Hypoproteinemia (Investigations) | 4 (7)
Hypoprotenemia (Investigations) | 1 (1)
Platelet Count Increased (Investigations) | 1 (2)
Platet Count Increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (21)
Dehydration (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (24)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (24)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 6 (21)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (9)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Arm Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (22)
Insomnia (Psychiatric disorders) | 1 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (5)
Skin Rash-Waist (Skin and subcutaneous tissue disorders) | 1 (4)
Skin rash-Waist (Skin and subcutaneous tissue disorders) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (4)
Bleeding at right injection site (Surgical and medical procedures) | 1 (1)
Soreness at injection site (Surgical and medical procedures) | 1 (1)
10020772-Hypertension (Vascular disorders) | 5 (20)
10021097-Hypotension (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03918499/Prot_SAP_000.pdf